CLINICAL TRIAL: NCT07042360
Title: Application of Comprehensive Non-invasive Assessment To Phenotype Tricuspid Regurgitation
Acronym: TRIREF
Status: Recruiting | Type: Observational
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr So Chak Yu kent, Clnincal assistant professor, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: 2025.229
Record Dates: First submitted 2025-06-06; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical treatment: Patient with >= moderate TR for medical treatment
  Interventions: Diagnostic Test: ReDs Pro; Diagnostic Test: Fibroscan
- Intervention: PAtient with >= moderate TR for transcather intervention
  Interventions: Diagnostic Test: ReDs Pro; Diagnostic Test: Fibroscan

INTERVENTIONS:
Diagnostic Test: ReDs Pro — The basic principle invovles emitting low-power electromagnetic sgnals into the lungs and measuring the dielectric properties of lung tissue
  The varing dielectric constants of these components result in differences in the impedance values for electromagnetic waves. Therefore, using the impedance method allows the estimation of the dielectric properties of lung tissue, which can be further converted into lung fluid content data through calculations.
Diagnostic Test: Fibroscan — Using external ultrasound scanner to check fo rliver stiffness using acoustic energy

SUMMARY:
Tricuspid regurgitation (TR) is an increasingly recognized valvular heart disease associated with high morbidity and mortality. With the availability of various novel transcatheter tricuspid interventions, it is no longer considered a "forgotten valve." Heart failure with preserved ejection fraction (HFpEF) is a prevalent condition also characterized by high morbidity and mortality. The prevalence of moderate to severe TR in the general population is 3% to 6%; however, in patients with heart failure (with reduced or preserved ejection fraction [EF]), the prevalence is 10% to 29%, rising to up to 39% in patients with HFpEF and atrial fibrillation (AF). The EuroTR registry, an international registry including patients who underwent percutaneous treatment for severe TR, reported that 72% of patients had a left ventricular ejection fraction (LVEF) ≥50%. In a subgroup of patients with right heart catheterization data, 68% had a pulmonary capillary wedge pressure (PCWP) ≥15 mm Hg, indicating that many of these patients may have HFpEF. Patients with significant TR have also been shown to experience irreversible liver derangement and cirrhosis. Non-invasive evaluation of liver stiffness (LS), measured by transient elastography, has recently received increased attention in patients with heart failure and has been shown to closely correlate with right-sided filling pressures. LS has been used to predict adverse outcomes in patients undergoing transcatheter aortic valve (TA) surgery with concomitant left-sided valve surgery.

On the other hand, the Remote Dielectric Sensing System (ReDS; Sensible Medical Innovations, Israel) is a device that measures lung fluid non-invasively and provides an objective and reproducible index of volume status. It is an FDAapproved device for heart failure patients. ReDS measurements are presented as the percentage of fluid relative to lung volume, with normal values ranging between 20% to 35%. Studies have demonstrated excellent correlations between the ReDS index and computed tomography (CT)-measured lung water and invasively determined hemodynamics. Additionally, it has been shown to predict heart failure rehospitalization in patients with acute heart failure.

Given the emergence of novel transcatheter tricuspid interventions and the established link between TR, HFpEF, and markers such as liver stiffness and lung fluid index (measured by ReDS), this study will examine the intricate interplay between these conditions and their shared pathophysiology. By analyzing left and right heart function, risk factors, and treatment outcomes, the research aims to phenotype TR using non-invasive assessment tools to predict clinical outcomes and improve treatment strategies for patients with different types of TR. Our findings will contribute to developing more effective and personalized treatment plans for patients with TR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with >=moderate TR
* able to consent for the study.

Exclusion Criteria:

1. LVEF <=40%
2. Have significant left sided organic valvular heart disease (i.e. >=moderate AS, >=moderate MS, >=moderate MR of organic or mixed aetiology), dysfunctional mitral valve replacement or aortic valve replacement
3. Prior tricuspid valve interventions (eg TriClip, tricuspid valve repair or replacement) (To allow accurate transient elastography)
4. Known hepatocellular carcinoma
5. Known portal vein thrombosis
6. Established liver cirrhosis with a known liver-related aetiology
7. Hepatitis C infection and not on treatment
8. Uncontrolled hepatitis (e.g. hepatitis B infection, autoimmune hepatitis)
9. Fatty liver with evidence of non-alcoholic fatty liver disease or cirrhosis (to allow accurate non-invasive lung fluid assessment)
10. recent rib fracture (<3 months) with or without flail chest
11. BMI <20 or >36
12. Height <155cm or >195cm
13. Patients with right lung tumor
14. Patients with right sided pacemaker
15. Patients with known underlying exudative right pleural effusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: By analyzing left and right heart function, risk factors, and treatment outcomes, the research aims to phenotype TR using non-invasive assessment tools to predict clinical outcomes and improve treatment strategies for patients with different types of TR.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Heart failure hospitalisation rate | 1 year
  Heart failure hospitalization rate of subjects at 1 year
Tricuspid valve intervention rate | 1 year
  Tricuspid valve intervention rate of subjects at 1 year
Cardiovascular mortality rate | 1 year
  Cardiovascular mortality rate of subjects at 1 year

SECONDARY OUTCOMES:
Heart failure hospitalisation rate | 6-month
  Heart failure hospitalization rate of subjects at 6-month
Tricuspid valve intervention rate | 12-month
  1-year tricuspid valve intervention of subjects at 12-month
NYHA Classification | 6-month
  Assess 6-month symptom burden via NYHA classification
NYHA Classification | 12-month
  Assess 1 year symptom burden via NYHA classification
Quality of Life measures | 6-month
  Assess Quality of Life measures of subject at 6-month via Kansas City Cardiomyophthy Questionnaire-12.
  Score range from 0-100, higher score indicates better outcome (Better Quality of Life/ less affected by Symptoms)
Quality of Life measures | 12-month
  Assess Quality of Life measures of subject at 12-month via Kansas City Cardiomyophthy Questionnaire-12 Score range from 0-100, higher score indicates better outcome (Better Quality of Life/ less affected by Symptoms)
Intensification of medical therapy | 6-month
  To monitor the short term use of intravenous diuretics at day-center at 6-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 6-month
  To monitor the increase of total daily dose oral diuretics at day-center at 6-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 6-month
  To monitor the short term use of inotrope at day-center at 6-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 6-month
  To monitor the application of aquapheresis at day-center at 6-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 12-month
  To monitor the short term use of intravenous diuretics at day-center at 12-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 12-month
  To monitor the increase of total daily dose oral diuretics at day-center at 12-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 12-month
  To monitor the short term use of inotrope at day-center at 12-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Intensification of medical therapy | 12-month
  To monitor the application of aquapheresis at day-center at 12-month follow-up to reflect if there is any intensification of medical therapy for treatment of Tricuspid Regurgitation
Echocardiographic parameters changes | 12-month
  Compare changes in TAPSE in patients at 12-months vs baseline using 3D Echocardiogram meaurements at 12-month follow up
Echocardiographic parameters changes | 12-month
  Compare changes in 3D Right Ventricle Ejection Fraction (RVEF) using 3D Echocardiogram meaurements in patients at 12-months vs baseline
Echocardiographic parameters changes | 12-month
  Compare changes in TAPSE/RVOT ratio in patients at 12-months vs baseline
Echocardiographic parameters changes | 12-month
  Compare changes in 3D RV volume in patients at 12-months vs baseline
Echocardiographic parameters changes | 12-month
  Compare changes in Right Ventricle size in patients at 12-months vs baseline using 3D Echocardiogram meaurements
Echocardiographic parameters changes | 12-month
  Compare changes in Right Ventricle Systolic Pressure (RVSP) in patients at 12-months vs baseline using 3D Echocardiogram meaurements at 12-month follow up
Echocardiographic parameters changes | 12-month
  Compare changes in Left ventricular ejection fraction (LVEF) in patients at 12-months vs baseline
Echocardiographic parameters changes | 12-month
  Compare changes in Left ventricular global longitudinal strain (LV GLS) in patients at 12-months vs baseline 8. 1 year worsening of left ventricular function (LVEF, GLS, LVOT VTI)
Intensification of medical therapy | 6-month
  6-month intensification of medical therapy of subjects (including short term use of intravenous diuretics at day-center, increase oral diuretics dose or frequency, short term use of inotrope at day-center, application of aquapheresis
Echocardiographic parameters changes | 12-month
  Compare changes in Left ventricular outflow tract (LVOT VTI) in patients at 12-months vs baseline using 3D Echocardiogram meaurements at 12-month follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Shatin, Hong Kong